CLINICAL TRIAL: NCT01276730
Title: A Pilot Phase II Two-Arm, Randomized Clinical Trial of Concomitant Immunotherapy (With Interferon-Alpha and Retinoic Acid) and Radiation Therapy for the Treatment of Advanced Cervical Cancer in India
Brief Title: Advanced Cervical Cancer Trial in India
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 464.05
Record Dates: First submitted 2010-11-02; First posted 2011-01-13 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Cervical Cancer
Keywords: Advanced cervical cancer; India
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Interferons; Tretinoin; Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Treatment consists of Interferon, given as a sub-cutaneous injection, 3 times per week for 4 weeks, 20 mg Retinoic Acid tablets, 2 times a day for 30 days. starting from the first day of radiation.
  Interventions: Drug: Interferon, Retinoic Acid and radiation
- Group B (Active Comparator): Treatment consists of radiation and chemotherapy using Cisplatin. Cisplatin, given intravenously, will be administered on the first day of each week, mixed with saline solution, before and after the Cisplatin infusion.
  Radiation will be given for a few minutes daily, five days a week, for approximately 5 weeks.
  Two weeks after completion of external radiotherapy, subject will receive internal radiation (brachytherapy) once a week for two weeks. For this internal radiation a specially designed instrument will be inserted into the vagina that will be connected to a machine for a few minutes.
  Interventions: Drug: Cisplatin and radiation

INTERVENTIONS:
Drug: Interferon, Retinoic Acid and radiation — Interferon-α2b will be administered 3 times a week for four weeks at a dose of 3 x 106 IU subcutaneously concomitant with radiotherapy. The first dose will be administered on the day the subject starts radiotherapy; 13-cis-retinoic acid will be administered orally at a dose of 40 mg/day for 1 month starting from day 1 of radiotherapy; a total of 40 to 45 Gy whole pelvis irradiation will be delivered in conventional fractions to both the study group and the control group. Additional parametrial dosages will be delivered to complete 55 Gy. This will be followed by two intracavitary applications of approximately 40-50 Gy, depending on the volume.
  Arms: Group A
Drug: Cisplatin and radiation — Weekly cisplatin will be administered concurrent with external beam radiation at a dose of 40mg/m2/week for 5 weeks; a total of 40 to 45 Gy whole pelvis irradiation will be delivered in conventional fractions. Additional parametrial dosages will be delivered to complete 55 Gy. This will be followed by two intracavitary applications of approximately 40-50 Gy, depending on the volume.
  Arms: Group B

SUMMARY:
The study objective:

* To evaluate the response and survival rates after treating stage III cervical cancer with retinoic acid and interferon-α combined with radiotherapy in the study group.
* To evaluate the response and survival rates after treating stage III cervical cancer patients with concomitant cisplatin and radiotherapy in the control group.
* To evaluate the safety and tolerability of the combination of retinoic acid, interferon-α and radiation therapy compared with concomitant chemo-radiation therapy.
* To determine if there is an immune response to Human Papillomavirus (HPV) by estimating serum IgG1 and IgG2 antibodies against E7 proteins of HPV types 16 and 18 before and after treatment.

The study hypothesis:

* The response rates and survival rates of retinoic acid and interferon-α combination with radiation will be better than chemo-radiation to treat stage III cervical cancer.
* Treatment with the retinoic acid, interferon-α and radiation combination therapy will be less toxic and better tolerated than chemo-radiation therapy.

DETAILED DESCRIPTION:
A total of 200 women with confirmed diagnosis of invasive cervical cancer, stage III, will be recruited into the study. The patients will be recruited from the Gynecologic Oncology Department of the Chittaranjan National Cancer Institute that registers more than 600 cases of cancer of the cervix per year. Computer-generated numbers will randomize patients into the two treatment arms.

This trial is designed to treat stage III cervical cancer patients with concomitant immunotherapy (with cis-retinoic acid and interferon-α) and radiotherapy in the study arm.

Cancer of the uterine cervix is the second most common cancer among women worldwide and is the cause of the largest number of cancer-related deaths among women in the developing countries. In India, cervical cancer is the commonest cancer among women (126,000 new cases, 71,000 deaths in 2000), accounting for more than a quarter of the global burden of cervical cancer (471,000 new cases and 233,000 deaths).1,2 In contrast, in the U.S., although, there were only 12,200 new cases of cervical cancer and 4,100 deaths in 2003, the United States spends $5 billion per year screening and treating cervical cancer and precancerous lesions.

Advanced cervical cancer is relatively rare in the developed world because of routine PAP testing. However, in a developing country like India, because of the absence of any population based cervical cancer screening programs (HPV testing, PAP smears), nearly 80% of the patients are initially detected at stage III or higher. Cisplatin-based chemotherapy administered along with surgery and radiation is the recommended treatment for advanced cervical cancer in the US and other developed countries.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cervical cancer

Exclusion Criteria:

* Previously treated for cancer of the cervix
* Karnofsky Performance Score less than 50
* Renal dysfunction ( Serum creatinine > 2.0mg/dl)
* Hepatic dysfunction (Serum bilirubin> 2.0 mg/dl, transaminases > 1.5 times normal)
* Pregnant or lactating women: Women will be tested by pregnancy test for possibility of existing pregnancy. Those that meet criteria of trial will be asked to promise that they don't become pregnant; barrier contraception will be recommended.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2007-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years or death
  Overall survival curves will be computed using the method of Kaplan and Meyer. The difference in survival between the two groups will be compared by log rank test with the O'Brien-Fleming boundaries to control for alpha spending at a planned interim analysis (50% of the total accrual).

SECONDARY OUTCOMES:
Response rate | 3 years or death
  Response rate will be compared between the arms. Response will be determined by radiological imaging and defined to include Complete Response, the disappearance of all gross evidence of disease, and Partial Response, more than 50% reduction in the two largest dimensions of the measurable tumor.
Overall toxicity | 3 years or death
  Fisher's exact test will be used to compare the incidences of WHO toxicities and response rates between the treatment groups.
Determine immune response to Human Papillomavirus HPV | 3 years to death
  By estimating serum IgGl and IgG2 antibodies against E7 protein of HPV types 16 and 18 before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Partha S Basu, MD, Principal Investigator — Chittaranjan National Cancer Institute
Locations (1):
- Chittaranjan National Cancer Institute, Kolkata, India

REFERENCES:
- [Derived] Basu P, Jenson AB, Majhi T, Choudhury P, Mandal R, Banerjee D, Biswas J, Pan J, Rai SN, Ghim SJ, Miller D. Phase 2 Randomized Controlled Trial of Radiation Therapy Plus Concurrent Interferon-Alpha and Retinoic Acid Versus Cisplatin for Stage III Cervical Carcinoma. Int J Radiat Oncol Biol Phys. 2016 Jan 1;94(1):102-110. doi: 10.1016/j.ijrobp.2015.09.040. PMID 26700705